CLINICAL TRIAL: NCT05884086
Title: Ataxia GAA-FGF14 - Descriptive Genetic and Clinical Study on Late Onset Ataxia Related to a GAA Expansion in the FGF14 Gene
Brief Title: Ataxia GAA-FGF14 - Descriptive Genetic and Clinical Study
Acronym: GAA-FGF14
Status: Active, not recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENAUD Mathilde, MD,PhD, Central Hospital, Nancy, France
Other Study IDs: 2023PI013-372
Record Dates: First submitted 2023-05-16; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Ataxia, Gait
Keywords: ataxia; spinocerebellar ataxia; genetic ataxia
MeSH Terms: conditions — Gait Ataxia; Ataxia; Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — no intervention is necessary. Clinical observation and clinical examination only.

SUMMARY:
Cerebellar ataxias of late onset are of undetermined etiology in many cases. A new cause of late-onset cerebellar ataxia was discovered in January 2023 corresponding to an expansion of GAA triplets in intron 1 of the FGF14 gene.

However, this cerebellar ataxia is still poorly known and requires further investigations to know its clinical phenotype and its evolution in order to propose a diagnosis and a genetic counseling adapted to patients and families. The objective of our study will be to describe the clinical and genotypic phenotype of patients with GAA-FGF14

DETAILED DESCRIPTION:
The objective of our study will be to describe the clinical and genotypic phenotype of patients with GAA-FGF14. We wish to describe the precise clinical phenotype by detailing each patient's clinical examination, medical history, treatment history, frequency and symptomatology of episodes, MRI radiological data, otho-rihno-laryngeal examination data etc . We would also like to describe the precise genotype for each patient, specifying the number of GAA expansions and its characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cerebellar ataxia of type GAA-FGF14

Exclusion Criteria:

* patients not wishing to be followed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of cerebellar ataxia of type GAA-FGF14 followed at the CHRU of Nancy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
description of clinical symptoms | through study completion, an average of 3 years
  description of clinical symptoms such as gait impairment, diplopia, vertigo, dizziness etc.
description of genotype | through study completion, an average of 3 years
  genotypic characterization of the GAA expansion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier régional universitaire, Nancy, France

REFERENCES:
- [Background] Pellerin D, Danzi MC, Wilke C, Renaud M, Fazal S, Dicaire MJ, Scriba CK, Ashton C, Yanick C, Beijer D, Rebelo A, Rocca C, Jaunmuktane Z, Sonnen JA, Lariviere R, Genis D, Molina Porcel L, Choquet K, Sakalla R, Provost S, Robertson R, Allard-Chamard X, Tetreault M, Reiling SJ, Nagy S, Nishadham V, Purushottam M, Vengalil S, Bardhan M, Nalini A, Chen Z, Mathieu J, Massie R, Chalk CH, Lafontaine AL, Evoy F, Rioux MF, Ragoussis J, Boycott KM, Dube MP, Duquette A, Houlden H, Ravenscroft G, Laing NG, Lamont PJ, Saporta MA, Schule R, Schols L, La Piana R, Synofzik M, Zuchner S, Brais B. Deep Intronic FGF14 GAA Repeat Expansion in Late-Onset Cerebellar Ataxia. N Engl J Med. 2023 Jan 12;388(2):128-141. doi: 10.1056/NEJMoa2207406. Epub 2022 Dec 14. PMID 36516086